CLINICAL TRIAL: NCT00839423
Title: Double-blind, Randomised, Placebo-controlled Study Comparing the Efficacy and Safety of Two Fixed Dosages of a Novel Antidepressant Compound to That of Placebo in Patients With Major Depressive Disorder
Brief Title: Randomised Placebo-controlled Venlafaxine-referenced Study of Efficacy and Safety of 5 and 10 mg of Vortioxetine (Lu AA21004) in Acute Treatment of Major Depressive Disorder in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11492A; 2006-001515-29 (EudraCT Number)
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Placebo-controlled; Active reference; Multicenter study; Randomised study; Acute treatment
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Vortioxetine (Lu AA21004) 5 mg (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)
- Vortioxetine (Lu AA21004) 10 mg (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)
- Venlafaxine XL 225 mg (Other): Active Reference
  Interventions: Drug: Venlafaxine XL

INTERVENTIONS:
Drug: Placebo — capsules, daily, orally
  Arms: Placebo
Drug: Vortioxetine (Lu AA21004) — encapsulated tablets, daily, orally
  Other Names: Brintellix
  Arms: Vortioxetine (Lu AA21004) 10 mg; Vortioxetine (Lu AA21004) 5 mg
Drug: Venlafaxine XL — capsules, daily, orally
  Other Names: Effexor®
  Arms: Venlafaxine XL 225 mg

SUMMARY:
The purpose of this Venlafaxine-referenced study is to evaluate the efficacy, safety and tolerability of two fixed doses of Vortioxetine in the acute treatment of Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* MDE as primary diagnosis according to DSM-IV-TR criteria (classification code 296.xx)
* Current MDE duration of at least 3 months and less than 12 months
* The patient has a MADRS total score >=30

Exclusion Criteria:

* Any current psychiatric disorder other than MDD as defined in the DSM-IV TR
* Any substance disorder within the previous 6 months
* Female patients of childbearing potential who are not using effective contraception
* Use of any psychoactive medication 2 weeks prior to screening and during the study

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Result] Alvarez E, Perez V, Dragheim M, Loft H, Artigas F. A double-blind, randomized, placebo-controlled, active reference study of Lu AA21004 in patients with major depressive disorder. Int J Neuropsychopharmacol. 2012 Jun;15(5):589-600. doi: 10.1017/S1461145711001027. Epub 2011 Jul 18. PMID 21767441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatients with Major Depressive Episode (MDE) were recruited from psychiatric settings.
Pre-assignment Details: Eligible patients were randomised equally (1:1:1:1) to one of the 4 treatment arms for a 6-week double-blind treatment period. The doses of Vortioxetine were 5 mg/day or 10 mg/day for 6 weeks. The dose of venlafaxine was 75 mg/day for 4 days, 150 mg/day for the following 3 days, and 225 mg/day for the remainder of the treatment period.
Groups:
- Vortioxetine 5 mg; Vortioxetine 10 mg: encapsulated tablets, daily, orally
- Venlafaxine 225 mg: capsules, daily, orally
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Venlafaxine 225 mg
Started | 105 | 108 | 100 | 113
Completed | 87 | 98 | 82 | 93
Not Completed | 18 | 10 | 18 | 20
Not completed — Adverse Event | 4 | 3 | 7 | 16
Not completed — Lack of Efficacy | 6 | 6 | 3 | 2
Not completed — Non-compliance | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 2 | 0
Not completed — Withdrawal of consent | 4 | 0 | 4 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Administrative or other reasons | 3 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Venlafaxine 225 mg | Total
Number analyzed (Participants) | 105 | 108 | 100 | 113 | 426
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (10.9) | 43.8 (11.6) | 42.3 (13.1) | 45.0 (10.3) | 43.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 70 | 66 | 62 | 267
  Male | 36 | 38 | 34 | 51 | 159
MADRS: Baseline Total Score [Mean (Standard Deviation); unit: units on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
  units on a scale | 33.9 (2.7) | 34.1 (2.6) | 34.0 (2.8) | 34.2 (3.1) | 34.0 (2.8)
Baseline 24-item HAM-D Total Score [Mean (Standard Deviation); unit: units on a scale] — The 24-item Hamilton Depression Rating Scale (HAM-D) is based on the 21-item HAM-D plus an additional 3 items (helplessness, hopelessness, and worthlessness). The observer makes his/her assessment on the basis of a specific statement, content, tone, facial expression, and gestures of the patient during the interview, and scores each item from 0 to 2 or 0 to 4. Total score from 0 to 76. The higher the score, the more severe.
  units on a scale | 29.7 (5.0) | 29.9 (5.4) | 29.3 (5.6) | 29.4 (5.0) | 29.6 (5.2)
HAM-A: Baseline Total Score [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56. The higher the score, the more severe.
  units on a scale | 22.9 (5.9) | 21.7 (6.2) | 22.3 (5.6) | 22.0 (5.5) | 22.2 (5.8)
CGI-S: Baseline Severity Score [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
  units on a scale | 5.1 (0.7) | 5.2 (0.7) | 5.1 (0.7) | 5.2 (0.7) | 5.2 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in MADRS Total Score After 6 Weeks of Treatment
Description: The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS) - all patients in the all-patients-treated set (APTS) who had at least one valid baseline and one valid post-baseline assessment of the MADRS total score; Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Venlafaxine 225 mg
Number analyzed (Participants) | 105 | 108 | 100 | 112
units on a scale | -14.50 (1.03) | -20.40 (1.01) | -20.20 (1.04) | -20.92 (0.99)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; The statistical model was an analysis of covariance (ANCOVA) of the change from baseline in MADRS total score (FAS, LOCF) with treatment and centre as fixed factors and the baseline MADRS score as a covariate. Null hypothesis: No difference between 10 mg Vortioxetine and placebo at Week 6. With 96 patients in each treatment arm and a standard deviation of 9 points, the power to detect a true effect of 3.7 points on the MADRS total score at Week 6 will be 80%; Test type: Superiority or Other; p < 0.0001, ANCOVA — A hierarchical hypothesis testing procedure was used. The comparison of 10 mg to placebo was primary. Since p-value was <0.05, hierarchically testing continued; Mean Difference (Final Values) = -5.70, 95% CI 2-sided [-8.49 to -2.91], Standard Error of Mean 1.42
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 5 mg; The statistical model was ANCOVA of the change from baseline in MADRS total score (FAS, LOCF) with treatment and centre as fixed factors and the baseline MADRS score as a covariate. Null hypothesis: No difference between 5 mg Vortioxetine and placebo at Week 6; Test type: Superiority or Other; p < 0.0001, ANCOVA — The hierarchical hypothesis testing meant that comparison of 5 mg to placebo was performed at a 5% significance level since significance was achieved for the primary comparison of 10 mg to placebo. Since p-value <0.05, hierarchically testing contd; Mean Difference (Final Values) = -5.90, 95% CI 2-sided [-8.64 to -3.17], Standard Error of Mean 1.39
Statistical Analysis 3: Comparison: Placebo vs Venlafaxine 225 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — This treatment arm was not in the testing sequence. A nominal p-value is provided; Mean Difference (Final Values) = -6.42, 95% CI 2-sided [-9.13 to -3.72], Standard Error of Mean 1.38

2. Secondary Outcome: Change From Baseline in MADRS Total Score After 1 Week of Treatment
Time Frame: Baseline and Week 1
Population: FAS, LOCF. Please note that 1 patient in each Vortioxetine group did not have a valid MADRS assessment at Week 1, but were included in the analysis because they had a valid MADRS assessment after Week 1.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Venlafaxine 225 mg
Number analyzed (Participants) | 105 | 107 | 99 | 112
units on a scale | -5.04 (0.50) | -5.26 (0.49) | -5.86 (0.51) | -4.50 (0.48)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; The statistical model was ANCOVA of the change from baseline in MADRS total score (FAS, LOCF) with treatment and centre as fixed factors and the baseline MADRS score as a covariate. Null hypothesis: No difference between 10 mg Vortioxetine and placebo at Week 1; Test type: Superiority or Other; p = 0.2377, ANCOVA — The hierarchical procedure meant that the above hypothesis was tested at a 5% significance level since significance was achieved for both 10 and 5 mg at Week 6. Since p-value was >0.05, hierarchically testing stopped here; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-2.17 to 0.54], Standard Error of Mean 0.69
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 5 mg; The statistical model was ANCOVA of the change from baseline in MADRS total score (FAS, LOCF) with treatment and centre as fixed factors and the baseline MADRS score as a covariate. Null hypothesis: No difference between 5 mg Vortioxetine and placebo at Week 1; Test type: Superiority or Other; p = 0.7489, ANCOVA — The hierarchical procedure meant that the above hypothesis was not tested since significance was not achieved for 10 mg at Week 1. A nominal p-value is provided; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-1.54 to 1.11], Standard Error of Mean 0.67
Statistical Analysis 3: Comparison: Placebo vs Venlafaxine 225 mg; Test type: Superiority or Other; p = 0.4142, ANCOVA — This treatment arm was not in the testing sequence. A nominal p-value is provided; Mean Difference (Final Values) = 0.54, 95% CI 2-sided [-0.77 to 1.85], Standard Error of Mean 0.67

3. Secondary Outcome: Change From Baseline in HAM-D 24 Total Score After 6 Weeks of Treatment
Description: The 24-item Hamilton Depression Rating Scale (HAM-D) is based on the 21-item HAM-D plus an additional 3 items (helplessness, hopelessness, and worthlessness). The observer makes his/her assessment on the basis of a specific statement, content, tone, facial expression, and gestures of the patient during the interview, and scores each item from 0 to 2 or 0 to 4. Total score from 0 to 76. The higher the score, the more severe.
Time Frame: Baseline and Week 6
Population: FAS, LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Venlafaxine 225 mg
Number analyzed (Participants) | 105 | 108 | 100 | 111
units on a scale | -12.23 (0.90) | -17.51 (0.89) | -17.57 (0.92) | -17.32 (0.88)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -5.28, 95% CI 2-sided [-7.69 to -2.88], Standard Error of Mean 1.22
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -5.33, 95% CI 2-sided [-7.79 to -2.88], Standard Error of Mean 1.25

4. Secondary Outcome: Change From Baseline in HAM-A Total Score After 6 Weeks of Treatment
Description: The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56. The higher the score, the more severe.
Time Frame: Baseline and Week 6
Population: FAS, LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Venlafaxine 225 mg
Number analyzed (Participants) | 101 | 102 | 95 | 106
units on a scale | -8.41 (0.74) | -11.71 (0.75) | -11.41 (0.77) | -11.29 (0.73)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.0011, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -3.30, 95% CI 2-sided [-5.27 to -1.33], Standard Error of Mean 1.00
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.0034, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -3.00, 95% CI 2-sided [-5.01 to -1.00], Standard Error of Mean 1.02

5. Secondary Outcome: Change From Baseline in CGI-S Score After 6 Weeks of Treatment
Description: The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
Time Frame: Baseline and Week 6
Population: FAS, LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Venlafaxine 225 mg
Number analyzed (Participants) | 105 | 108 | 100 | 111
units on a scale | -1.55 (0.14) | -2.45 (0.14) | -2.51 (0.15) | -2.58 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-1.28 to -0.52], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.34 to -0.56], Standard Error of Mean 0.20

6. Secondary Outcome: Change in Clinical Status Using CGI-I Score at Week 6
Description: The Clinical Global Impression - Global Improvement (CGI-I) is a 7-point scale rated from 1 (very much improved) to 7 (very much worse). The investigator rated the patient's overall improvement relative to baseline, whether or not, in the opinion of the investigator, this was entirely due to the drug treatment.
Time Frame: Week 6
Population: FAS, LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Venlafaxine 225 mg
Number analyzed (Participants) | 105 | 108 | 100 | 111
units on a scale | 2.64 (0.12) | 2.05 (0.12) | 2.04 (0.12) | 1.96 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.0003, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-0.90 to -0.27], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.0003, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-0.92 to -0.27], Standard Error of Mean 0.16

7. Secondary Outcome: Proportion of Responders at Week 6 (Response Defined as a >=50% Decrease in the MADRS Total Score From Baseline)
Time Frame: Week 6
Population: FAS, LOCF
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Venlafaxine 225 mg
Number analyzed (Participants) | 105 | 108 | 100 | 112
percentage of patients | 44.8 | 66.7 | 68.0 | 72.3
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.002, Fisher Exact — A nominal p-value is provided; Difference % = 21.90, 95% CI 2-sided [8.89 to 34.92]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.001, Fisher Exact — A nominal p-value is provided; Difference % = 23.34, 95% CI 2-sided [10.05 to 36.43]

8. Secondary Outcome: Proportion of Remitters at Week 6 (Remission is Defined as a MADRS Total Score <=10)
Time Frame: Week 6
Population: FAS, LOCF
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Venlafaxine 225 mg
Number analyzed (Participants) | 105 | 108 | 100 | 112
percentage of patients | 26.7 | 49.1 | 49.0 | 55.4
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.001, Fisher Exact — A nominal p-value is provided; Difference % = 22.41, 95% CI 2-sided [9.74 to 35.07]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.001, Fisher Exact — A nominal p-value is provided; Difference % = 22.33, 95% CI 2-sided [9.39 to 35.28]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: 6-week double-blind treatment period and 4-week safety follow-up period Other Adverse Events: 6-week double-blind treatment period
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Venlafaxine 225 mg
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/108 | 2/100 | 1/113
Other Adverse Events (participants affected / at risk) | 53/105 | 63/108 | 66/100 | 78/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=105) | Vortioxetine 5 mg (N=108) | Vortioxetine 10 mg (N=100) | Venlafaxine 225 mg (N=113)
Varicella (Infections and infestations) | 0 | 0 | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=105) | Vortioxetine 5 mg (N=108) | Vortioxetine 10 mg (N=100) | Venlafaxine 225 mg (N=113)
Vision blurred (Eye disorders) | 2 | 2 | 1 | 6
Constipation (Gastrointestinal disorders) | 1 | 1 | 3 | 11
Diarrhoea (Gastrointestinal disorders) | 5 | 9 | 7 | 5
Dry mouth (Gastrointestinal disorders) | 7 | 8 | 8 | 19
Nausea (Gastrointestinal disorders) | 10 | 32 | 38 | 38
Vomiting (Gastrointestinal disorders) | 1 | 2 | 9 | 4
Fatigue (General disorders) | 6 | 4 | 6 | 11
Nasopharyngitis (Infections and infestations) | 9 | 8 | 7 | 4
Dizziness (Nervous system disorders) | 8 | 7 | 7 | 14
Headache (Nervous system disorders) | 26 | 23 | 25 | 32
Tremor (Nervous system disorders) | 3 | 5 | 0 | 6
Anorgasmia (Psychiatric disorders) | 0 | 0 | 0 | 7
Insomnia (Psychiatric disorders) | 5 | 7 | 6 | 14
Ejaculation delayed (Reproductive system and breast disorders) | 0/36 | 0/38 | 0/34 | 4/51
Erectile dysfunction (Reproductive system and breast disorders) | 0/36 | 0/38 | 0/34 | 4/51
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 3 | 10 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The main publication has to be published before any sub publication. The investigators shall obtain Lundbeck's written approval before publishing any publication relating to Vortioxetine, the Study, the Protocol and/or the results recorded during the Study.